CLINICAL TRIAL: NCT02369289
Title: Bone Mineral Density in Israeli Female Vegans and Omnivores
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0013-15-TLV
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Bone Mineral Density; Vegan Diet
MeSH Terms: interventions — Bone Density

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- vegans: a vegan diet in the last 3 years
  Interventions: Other: bone mineral density test
- omnivores: aminal-based diet, comsumption of aminal products at least 3 times a week
  Interventions: Other: bone mineral density test

INTERVENTIONS:
Other: bone mineral density test

SUMMARY:
A vegan diet is more and more prevalent in the general population in Israel in recent years. There have been some concerens that a vegan diet may lack in bone-health related nutrients (such as calcium, protein and vitamin D), and therefore may cause a decreased bone mineral density. The study aims to compare bome mineral density and other biochemical bone health parameters in vegan and omnivore non-menopausal Israely females.

ELIGIBILITY:
Inclusion Criteria:

* generaly healthy
* vegan group: vegan diet for the past 3 years
* omnivore group: comsumption of animal products at least 3 times a week

Exclusion Criteria:

* pragnent / breastfeeding women
* amenorrhea (absence of a menstrual period) for more than 3 months
* amenorrhea in the past
* significant underweight in the present/past (BMI < 17.5)
* taking medicine that affect bone density
* hypo/hyper thyroidism
* hypo/hyper parathyroidism
* smokimg in the past 10 years
* over consumption of alcohol (more than 7 units a week)

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: generaly healthy vegan and omnivore females, age 30-45
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel